CLINICAL TRIAL: NCT02122120
Title: Home Enteral Nutrition (HEN) Reduces Complications, Length of Stay and Health-care Costs: Results From the Multicenter Study.
Brief Title: The Value of Aritficial Diet and Complex Care in Home Nutrition
Status: Completed | Type: Observational
Sponsor: Stanley Dudrick's Memorial Hospital (Other)
Responsible Party: Principal Investigator, Stanislaw Klek, Head of the Departement, Stanley Dudrick's Memorial Hospital
Other Study IDs: HEN1
Record Dates: First submitted 2014-04-19; First posted 2014-04-24 (Estimated); Last update posted 2014-04-24 (Estimated); Status verified 2014-04

CONDITIONS: Dietary Modification
Keywords: enteral nutrition, tube feeding, nutritional support

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Before HEN: Patients with tube feeding with kitchen diet for at least twelve months
  Interventions: Dietary Supplement: HEN

INTERVENTIONS:
Dietary Supplement: HEN — Patients with tube feeding with FSMP for at least twelve months

SUMMARY:
Home enteral nutrition (HEN) has always been recognized as a life-saving procedure, but with the ongoing economic crisis influencing health care, its cost-effectiveness has been questioned recently.

Objective: The unique reimbursement situation in Poland enabled the otherwise ethically unacceptable, hence unavailable, comparison of the period of no-feeding and the long-term feeding and the subsequent analyses of the clinical value of the latter and its cost-effectiveness.

DETAILED DESCRIPTION:
Background: Home enteral nutrition (HEN) has always been recognized as a life-saving procedure, but with the ongoing economic crisis influencing health care, its cost-effectiveness has been questioned recently.

Objective: The unique reimbursement situation in Poland enabled the otherwise ethically unacceptable, hence unavailable, comparison of the period of no-feeding and the long-term feeding and the subsequent analyses of the clinical value of the latter and its cost-effectiveness.

Design: The observational multicentre study in the group of 456 HEN patients was performed between January 2007 and July 2013. Two twelve-month periods were compared. During the first one patients were tube fed with home-made diet without monitoring, while during the other the complex HEN was carried out. The latter included tube feeding and complex monitoring by nutrition support team. Number of complications, hospital admissions, length of hospital stay (LOS), biochemical and anthropometric parameters and costs of hospitalization were compared.

ELIGIBILITY:
Inclusion Criteria:

* indications for home tube feeding (HTF),
* complete present and past medical history,
* tube feeding for at least twelve months before HEN and at least twelve months afterwards.

Exclusion Criteria:

* doubtful indications for HEN, no access or an incomplete medical record,
* treatment period shorter than 12 months either before or after enrolment

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: 456 patients during home tube feeding
Sampling Method: Probability Sample
Enrollment: 456 (Actual)
Dates: Start 2007-01; Primary Completion 2012-12 (Actual); Study Completion 2013-01 (Actual)

PRIMARY OUTCOMES:
Number of complications | 24 moths

SECONDARY OUTCOMES:
Number of hospital admissions | 24 months

OTHER OUTCOMES:
length of hospital stay | 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Stanislaw Klek, MD PhD, Principal Investigator — Stanley Dudrick's Memorial Hospital
Locations (1):
- Stanley Dudrick's Memorial Hospital, Skawina, Malopolska, Poland

REFERENCES:
- [Background] Majka AJ, Wang Z, Schmitz KR, Niesen CR, Larsen RA, Kinsey GC, Murad AL, Prokop LJ, Murad MH. Care coordination to enhance management of long-term enteral tube feeding: a systematic review and meta-analysis. JPEN J Parenter Enteral Nutr. 2014 Jan;38(1):40-52. doi: 10.1177/0148607113482000. Epub 2013 Mar 25. PMID 23528323
- [Derived] Klek S, Hermanowicz A, Dziwiszek G, Matysiak K, Szczepanek K, Szybinski P, Galas A. Home enteral nutrition reduces complications, length of stay, and health care costs: results from a multicenter study. Am J Clin Nutr. 2014 Aug;100(2):609-15. doi: 10.3945/ajcn.113.082842. Epub 2014 Jun 25. PMID 24965306